CLINICAL TRIAL: NCT06200870
Title: Iron Deficiency as a Promoter of Intra-leaflet Haemorrhage-induced Aortic Valve Calcification
Brief Title: ID as a Promoter of IH-induced CAVD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Chuanbao Li, Prof., Qilu Hospital of Shandong University
Other Study IDs: 2023IDCAVD-LCB
Record Dates: First submitted 2023-11-05; First posted 2024-01-11 (Actual); Last update posted 2024-01-11 (Actual); Status verified 2023-12

CONDITIONS: Iron Deficiencies; Calcified Aortic Valve
MeSH Terms: conditions — Iron Deficiencies; Aortic Valve, Calcification of

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- aortic valvular sclerosis group
- non-aortic valvular sclerosis group

SUMMARY:
Calcific aortic valve disease (CAVD) is a highly prevalent, disabling and costly disorder with generally poor long-time outcomes once critical stenosis presents with symptoms. Elucidating viable therapeutic strategies for CAVD is pressing. Valvular interstitial cells (VICs) control the structure and function of aortic valve. Intra-leaflet haemorrhage (IH), commonly occurring in histologically stenotic aortic valves, while, in 2019, researchers pointed that iron deposits also presented obviously healthy valves. In line with this, later exploration from vitro showed that iron stimulation alone could not promote VICs calcification. Iron deficiency (ID) is a frequent co-morbidity in multiple chronic cardiovascular diseases such as CAVD; up to 50% of patients with severe aortic stenosis present ID. Data from a small clinical study in patients undergoing TAVI showed those in ID status appeared much higher mean transaortic gradient; whereas no studies have assessed the correlation between ID and aortic valve remodelling and dysfunction progress itself. Here, the investigators aim to investigate for a tentative correlation between ID and human aortic valve remodeling and dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* if performed with both color doppler echocardiography and anemia profile on admission as part of routine checkup.

Exclusion Criteria:

* if younger than the age of 18;
* if no anemia profile or doppler echocardiography was measured;
* if anemia profile or doppler echocardiography was analyzed in external laboratories;
* if had a history of rheumatic heart disease, infective endocarditis or any other congenital disorders that may implicate aortic valve structures, such as bicuspid aortic valve morphology, Marfan syndrome, and so on.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients at the outpatient clinic or inpatient department, Qilu hospital of Shandong University, Jinan, were recruited during the period from January 2018 to March 2023.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Serum iron | within 24 hours of admission
  Plasma levels of serum iron will be reported in μmol/L.
Total iron binding capacity | within 24 hours of admission
  Total iron binding capacity will be reported in μmol/L.
Serum transferrin receptor | within 24 hours of admission
  Plasma levels of serum transferrin receptor will be reported in g/L.
Unsaturated iron-binding capacity | within 24 hours of admission
  Serum iron and total iron binding capacity will be combined to report unsaturated iron-binding capacity in μmol/L.
Serum transferrin | within 24 hours of admission
  Plasma levels of serum transferrin will be reported in g/L.
Transferrin saturation | within 24 hours of admission
  Serum iron and total iron binding capacity will be combined to report transferrin saturation in %.
Soluble transferrin index | within 24 hours of admission
  Serum iron and serum transferrin will be combined to report soluble transferrin index.

IPD SHARING:
Plan to Share IPD: No
Limited by the submitted ethical protocols